CLINICAL TRIAL: NCT02363270
Title: Comparison of Intravenous Push Dose of Low Dose Ketamine to Short Infusion of Low Dose Ketamine for Treatment of Moderate to Severe Pain in the Emergency Department: A Prospective, Randomized, Double-Blind Study
Brief Title: Ketamine: Comparison of IV Push vs. IV Drip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Manager, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-10-08-MMC
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-10

CONDITIONS: Pain
Keywords: Analgesia; ketamine
MeSH Terms: conditions — Pain; Agnosia | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV Push Group (Active Comparator): Ketamine medication given via IV Push. IV Push is the intervention.
  Interventions: Procedure: Ketamine
- IV Drip Group (Active Comparator): Ketamine medication given via IV Drip. IV Drip is the intervention.
  Interventions: Procedure: Ketamine

INTERVENTIONS:
Procedure: Ketamine — IV Push or or IV Drip

SUMMARY:
Our previous published research comparing the efficacy of intravenous ketamine to morphine has shown ketamine to provide equivalent relief of moderate to severe acute pain in emergency medicine patients. Secondary analysis of the previous published research has also revealed ketamine to have statistically more side effects. The investigators believe that increasing the time of administration of the ketamine, from a push injection to a drip infusion, will minimize the side effects experienced by recipients of ketamine.

DETAILED DESCRIPTION:
Ketamine is a noncompetitive N-methyl D-aspartate (NMDA) receptor antagonist that blocks the release of excitatory neurotransmitter glutamate and provides anesthesia, amnesia and analgesia by virtue of decreasing central sensitization and "wind-up" phenomenon. At low (sub-dissociative, analgesics) doses of 0.1-0.4 mg/kg either as an adjunct to opioid analgesics or as a single agent, ketamine provides good analgesia while preserving airway patency, ventilation, and cardiovascular stability. In addition, the low-dose of ketamine increases the analgesic potency of opioids thus decreasing their requirements. Several recent studies of low-dose ketamine administered together with morphine provided acceptable pain relief to 55-60% of patients with minor side effects of dizziness, nausea and feeling of unreality. More recently the investigators conducted a research comparing Low-Dose Ketamine to Morphine for Moderate to Severe Pain in the Emergency Department with respect its analgesic efficacy and safety. Results demonstrated similar pain relief at 30 min between 2 groups. However, 70% of patients in ketamine group had minor side effects at 5 min and 35% of patients at 30 min, as compared to 51% at 5 min. and 31% at 15 min. in the morphine group. The most common side effects reported by ketamine patients were dizziness, nausea, feeling of unreality, and mood changes.

Based on the above mentioned data from our previous published research study, we hypothesized that low-dose ketamine given as a short infusion over 15 min will provide similar analgesic efficacy as an intravenous push-dose but with much less side effects. There are several research papers that support our hypothesis.

A prospective, randomized trial compared two analgesic regimens, morphine with ketamine (K group) or morphine with placebo (P group) for severe acute pain in 73 trauma patients with a visual analog scale (VAS) score of at least 60/100. Morphine was administered at 0.1mg/kg and patients in the K group received 0.2 mg/kg of intravenous ketamine over 10 minutes, and the patients in the P group received isotonic sodium chloride solution. The results showed comparable change in VAS score at 30 minutes (34 mm (K) vs. 39 mm (P)) but reduced morphine consumption in the ketamine group (0.14 mg/kg (K) vs 0.2 mg/kg (P)).

A double-blind trial of 40 adult patients with acute musculoskeletal trauma compared a low-dose ketamine by subcutaneous infusion (0.1 mg/kg/h) with intermittent morphine (0.1 mg/kg IV every 4 hours ) and demonstrated better pain relief, less sedation and less nausea and vomiting with ketamine infusion than with intermittent morphine. In addition, none of the patients in ketamine group required supplementary analgesia.

A prospective case series of 20 unselected adult ED patients with acute pain that evaluated analgesic feasibility of low-dose ketamine infusion was conducted in an urban public hospital over a course of 5 months. Patients received 15mg of intravenous push dose ketamine that was followed by continuous ketamine infusion at 20mg per hour for one hour. Optional morphine (4 mg) was offered at 20, 40 and 60 minutes. Pain intensity was assessed at regular intervals for 2 hours using a 10-point verbal numerical rating scale (NRS), along with vital signs and levels of sedation. Results showed that fifteen patients reported clinically significant pain relief at 60 minutes and 13 at 120 minutes; and eighteen patients reported mild or modest side effects including dizziness, fatigue and headache.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Medicine patients
* Adult patients (18-65 years of age)
* Moderate to severe pain (Numeric Pain Rating Score =5).
* Patients must be awake, alert and oriented to time, place and person.
* Patients must be able to demonstrate understanding of the informed consent, and also able to verbalize how much pain they are having on the 10 point Numeric Rating Pain Scale, and the nature of the side effects they may be experiencing from the IV analgesia

Exclusion Criteria:

* Patients with cognitive deficits that are not able to demonstrate understanding as described above.
* Patient's reported weight of less than 45kg or more than 115kg.
* Patients with altered mental status, alcohol intoxication, eye trauma.
* Patients with hemodynamic instability (Systolic Blood pressure <90), and malignant hypertension.
* allergy to ketamine
* Pregnancy or breast feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2016-08-15 (Actual); Study Completion 2017-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Motov, MD, Principal Investigator — Maimonides Medical Center; John Marshall, MD, Study Chair — Maimonides Medical Center; Christian Fromm, MD, Study Director — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. Abdullah M. Ketamine. A new look at an old drug. M ABDULLAH. anaesthetics.ukzn.ac.za/.../Ketamine_a_new_look_at_an_old_drug_...(accessed on 12/21/11)
- [Background] Javery KB, Ussery TW, Steger HG, Colclough GW. Comparison of morphine and morphine with ketamine for postoperative analgesia. Can J Anaesth. 1996 Mar;43(3):212-5. doi: 10.1007/BF03011736. PMID 8829857
- [Background] Lester L, Braude DA, Niles C, Crandall CS. Low-dose ketamine for analgesia in the ED: a retrospective case series. Am J Emerg Med. 2010 Sep;28(7):820-7. doi: 10.1016/j.ajem.2009.07.023. Epub 2010 Apr 2. PMID 20837262
- [Background] Richards JR, Rockford RE. Low-dose ketamine analgesia: patient and physician experience in the ED. Am J Emerg Med. 2013 Feb;31(2):390-4. doi: 10.1016/j.ajem.2012.07.027. Epub 2012 Oct 4. PMID 23041484
- [Background] Gurnani A, Sharma PK, Rautela RS, Bhattacharya A. Analgesia for acute musculoskeletal trauma: low-dose subcutaneous infusion of ketamine. Anaesth Intensive Care. 1996 Feb;24(1):32-6. doi: 10.1177/0310057X9602400106. PMID 8669651
- [Background] Galinski M, Dolveck F, Combes X, Limoges V, Smail N, Pommier V, Templier F, Catineau J, Lapostolle F, Adnet F. Management of severe acute pain in emergency settings: ketamine reduces morphine consumption. Am J Emerg Med. 2007 May;25(4):385-90. doi: 10.1016/j.ajem.2006.11.016. PMID 17499654
- [Background] Ahern TL, Herring AA, Miller S, Frazee BW. Low-Dose Ketamine Infusion for Emergency Department Patients with Severe Pain. Pain Med. 2015 Jul;16(7):1402-9. doi: 10.1111/pme.12705. Epub 2015 Feb 3. PMID 25643741

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IV Push Group | IV Drip Group
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Push Group | IV Drip Group | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 48
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.25 (15.12) | 43.56 (12.32) | 44.40 (13.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 9 | 12 | 21
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Overall Rate of Feeling Unreality
Description: Overall rate of feeling of unreality as measured by Side Effects Rating Scale for Dissociative Anesthetics (SERSDA)
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | IV Push Group | IV Drip Group
Number analyzed (Participants) | 24 | 24
Participants | 22 | 13

ADVERSE EVENTS:
Time Frame: 120 minutes
Arm/Group | IV Push Group | IV Drip Group
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 22/24 | 13/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IV Push Group (N=24) | IV Drip Group (N=24)
Feeling of Unreality (Nervous system disorders) | 22 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No